CLINICAL TRIAL: NCT05921825
Title: Red Cell Distribution Width and Lactate Albumin Ratio as Prognostic Markers for Mortality in Sepsis and Septic Shock Patients
Brief Title: Red Cell Distribution Width and Lactate Albumin Ratio as Prognostic Markers for Mortality in Sepsis and Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shimaa Saad Mohamed Awd, Assistant lecturer, Tanta University
Other Study IDs: 34640/4/12
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Morality; Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Erythrocyte Indices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non survivors group: At 28 day, patients were divided into Non survivors group and Survivors group.
  Interventions: Diagnostic Test: Red cell distribution width; Diagnostic Test: lactate albumin ratio measurement
- Survivors group: At 28 day, patients were divided into Non survivors group and Survivors group.
  Interventions: Diagnostic Test: Red cell distribution width; Diagnostic Test: lactate albumin ratio measurement

INTERVENTIONS:
Diagnostic Test: Red cell distribution width — Blood will be drawn from the peripheral vein, arterial or a central catheter. This procedure will be done at diagnosis, 3 ,7, 14 and 21 days of sepsis
Diagnostic Test: lactate albumin ratio measurement — Blood will be drawn from the peripheral vein, arterial or a central catheter. This procedure will be done at diagnosis, 3 ,7, 14 and 21 days of sepsis

SUMMARY:
The aim of this study is to find the utility of red cell distribution width and lactate/albumin ratio as prognostic markers in sepsis and septic shock patients.

DETAILED DESCRIPTION:
Several indicators are being used to predict the prognosis of sepsis. Commonly used prognostic indicators include Acute Physiological and chronic health evaluation II (APACHE II), Sequential Organ Failure Assessment (SOFA), Mortality in Emergency Department Score (MEDS), New York Sepsis severity score.

Red cell distribution Width and lactate albumin ratio are being investigated for there prognostic value in septic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 60 years old.
2. Clinical criteria of sepsis
3. Or clinical criteria of septic shock including sepsis with persisting hypotension requiring vasopressors to maintain mean arterial pressure > 65 mmHg and having a serum lactate level > 2 mmol/L despite adequate volume resuscitation.

Exclusion Criteria:

1. No informed consent.
2. Patient with incomplete information and data.
3. The patient who received blood transfusion within 90 days before emergency admission.
4. The patients who are known to have long-term conditions causing anemia like sickle cell anemia, thalassemia, iron deficiency anemia.
5. Malignancy and chemotherapy during the previous 90 days.
6. Patients with either hepatic dysfunction, renal failure, having any disease in which albumin should be supplemented as liver cirrhosis with ascites, nephrotic syndrome and burns.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients of both sex with age between (18:60) years old admitted to surgical intensive care unit suffering from sepsis or septic shock will be enrolled in the study after fulfillments of inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
The prediction of mortality | 28 days
  The diagnostic accuracy for prediction of 28th day mortality by Red cell distribution Width and lactate albumin ratio.

SECONDARY OUTCOMES:
Length of intensive care stay | 28 days or till discharge from intensive care.
  Length of intensive care stay from admission till discharge either to the ward or mortality.
Extent of organ dysfunctions in patients with severe sepsis and septic shock | 28 days
  Organ dysfunction can be confirmed by acute change in sepsis-related organ failure assessment (SOFA).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author from one year after study completion
Supporting Information: Study Protocol
Time Frame: From one year after study completion
Access Criteria: The data will be available upon reasonable request from the corresponding author